CLINICAL TRIAL: NCT05304663
Title: A Study to Evaluate the Safety and Efficacy of Different Administration Sequences of L19TNF in Combination With Lomustine in Patients With Glioblastoma at First Progression
Brief Title: Safety and Efficacy of Different Administration Sequences of L19TNF With Lomustine in Glioblastoma at First Progression
Acronym: GLIOASTRA
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The Sponsor had no further plan for the study in object
Sponsor: Philogen S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PH-L19TNFLOM-05/21
Record Dates: First submitted 2022-02-24; First posted 2022-03-31 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Lomustine

STUDY DESIGN:
Intervention Model Description: Open label phase I study in subjects with glioblastoma at first progression to explore two different administration schedules of lomustine for the combination with L19TNF (ARM 1 and ARM 2).
  Patients will be assigned in an alternating fashion to ARM 1 or ARM 2 as long as both treatment arms are open. Should one treatment arm be stopped as more or equal to two dose limiting toxicities occur in this treatment arm, then all remaining patients will be assigned to the treatment arm that is still open until also this treatment arm will be stopped.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM 1: Fractionating Lomustine (Experimental): Patients will be treated in escalating cohorts of 6 patients with 10 µg/kg L19TNF on Days 1, 3 and 5, and on Days 22, 24 and 26 and lomustine at different doses on Day 1 and Day 22 (taken in the evening after L19TNF infusion) of a 42-day cycle for up to a maximum of 6 cycles.
  * Cohort 1: 10 µg/kg L19TNF and 60 mg/m2 lomustine
  * Cohort 2: 10 µg/kg L19TNF and 75 mg/m2 lomustine
  Interventions: Drug: Onfekafusp alfa; Drug: Lomustine
- ARM 2: Priming with L19TNF (Experimental): Patients will be treated in escalating cohorts of 6 patients with 10 µg/kg L19TNF on Days 1, 3 and 5, and on Days 22, 24 and 26 and lomustine at different doses on Day 5 (in the evening after infusion of L19TNF) of a 42-day cycle for up to a maximum of 6 cycles.
  * Cohort 1: 10 µg/kg L19TNF and 90 mg/m2 lomustine
  * Cohort 2: 10 µg/kg L19TNF and 110 mg/m2 lomustine In each arm, patients will be enrolled sequentially and no more than 2 patients will be treated in Cycle 1 in the same arm in parallel.
  Recruitment to an arm will be stopped should ≥ 2 DLTs occur in a cohort.
  Interventions: Drug: Onfekafusp alfa; Drug: Lomustine

INTERVENTIONS:
Drug: Onfekafusp alfa — Patients will be treated with 10 µg/kg L19TNF on Days 1, 3 and 5, and on Days 22, 24 and 26
  Other Names: L19TNF
Drug: Lomustine — Arm 1: Patients will be treated in escalating cohorts of 6 patients with lomustine at different doses (60 mg/m2 and 75 mg/m2) on Day 1 and Day 22 (taken in the evening after L19TNF infusion) of a 42-day cycle for up to a maximum of 6 cycles.
  Arm 2: Patients will be treated in escalating cohorts of 6 patients with lomustine at different doses (90 mg/m2 and 110 mg/m2) on Day 5 (in the evening after infusion of L19TNF) of a 42-day cycle for up to a maximum of 6 cycles.

SUMMARY:
Open label phase I study in subjects with glioblastoma at first progression to explore two different administration schedules of lomustine for the combination with L19TNF (ARM 1 and ARM 2).

Patients will be assigned in an alternating fashion to ARM 1 "Fractionating lomustine" or ARM 2 "Priming with L19TNF" as long as both treatment arms are open. Should one treatment arm be stopped as more or equal to two dose limiting toxicities occur in this treatment arm, then all remaining patients will be assigned to the treatment arm that is still open until also this treatment arm will be stopped.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥18.
2. Patients with histologically confirmed glioblastoma per 2021 WHO classification at first progression according to RANO criteria. Imaging data on progression must be available. Resection as previous treatment for progression or recurrence is allowed.
3. MGMT promotor methylation status known or tumor tissue for analysis available.
4. Presence of at least one lesion of measurable disease of 10 x 10 mm in longest perpendicular diameters on baseline MRI according to RANO criteria.
5. Karnofsky performance status (KPS) ≥ 60%.
6. Documented negative test for HIV-HBV-HCV. For HBV serology, the determination of HBsAg and anti-HBcAg Ab is required. In patients with serology documenting previous exposure to HBV, negative serum HBV-DNA is required. For HCV, HCV-RNA or HCV antibody test is required. Subjects with a positive test for HCV antibody but no detection of HCV-RNA indicating no current infection are eligible.
7. Female patients: female patients must be either documented not Women Of Childbearing Potential (WOCBP)* or must have a negative pregnancy test within 14 days of starting treatment. Additionally WOCBP must agree to use, from the screening to 6 months following the last study drug administration, highly effective contraception methods, as defined by the "Recommendations for contraception and pregnancy testing in clinical trials" issued by the Head of Medicine Agencies' Clinical Trial Facilitation Group (www.hma.eu/ctfg.html) and which include, for instance, progesterone-only or combined (estrogen- and progesterone-containing) hormonal contraception associated with inhibition of ovulation, intrauterine devices, intrauterine hormone-releasing systems, bilateral tubal occlusion or vasectomized partner.

   Male patients: male subjects able to father children must agree to use two acceptable methods of contraception throughout the study (e.g. condom with spermicidal gel). Double-barrier contraception is required.
8. Personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
9. Willingness and ability to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures.

   * Women of childbearing potential are defined as females who have experienced menarche, are not postmenopausal (12 months with no menses without an alternative medical cause) and are not permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral oophorectomy, or bilateral salpingectomy).

Exclusion Criteria:

1. Inability to undergo contrast-enhanced MRI.
2. Prior treatment for glioblastoma at recurrence, except surgery.
3. Surgical resection or biopsy of glioma within 4 weeks of the start of study treatment.
4. Previous treatment with L19TNF.
5. Known history of allergy to TNF or lomustine, any excipient in the study medication or any other intravenously administered human proteins/peptides/antibodies.
6. Absolute neutrophil count (ANC) < 1.5 x 10^9/L; platelets < 100 x 10^9/L or haemoglobin (Hb) < 9.0 g/dl.
7. Chronically impaired renal function as indicated by creatinine clearance < 60 mL/min or serum creatinine > 1.5 ULN.
8. Inadequate liver function (ALT, AST, ALP ≥ 2.5 x ULN or total bilirubin ≥ 2.0 x ULN).
9. INR > 1.5 ULN.
10. Any severe concomitant condition which makes it undesirable for the patient to participate in the study or which could jeopardize compliance with the protocol, in the opinion of the investigator.
11. Active or history of autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent, in the judgement of the investigator.
12. History within the last year of cerebrovascular disease and/or acute or subacute coronary syndromes including myocardial infarction, unstable or severe stable angina pectoris.
13. Heart insufficiency (> Grade II, New York Heart Association (NYHA) criteria).
14. Clinically significant cardiac arrhythmias or requiring permanent medication.
15. LVEF <55% or any other abnormalities observed during baseline ECG and echocardiogram investigations that are considered as clinically significant by the investigator. Subjects with current or a history of QT/QTc prolongation are excluded.
16. Uncontrolled hypertension.
17. Known arterial aneurism at high risk of rupture.
18. Ischemic peripheral vascular disease (Grade IIb-IV according to Leriche-Fontaine classification).
19. Anxiety ≥ CTCAE Grade 3.
20. Severe diabetic retinopathy such as severe non-proliferative retinopathy and proliferative retinopathy.
21. Major trauma including major surgery (such as abdominal/cardiac/thoracic surgery) within 3 weeks of administration of study treatment.
22. Known history of tuberculosis.
23. Pregnancy or breast feeding.
24. Requirement of chronic administration of high dose corticosteroids or other immunosuppressant drugs. Subjects must have been either off corticosteroids, or on a stable or decreasing dose ≤ 4 mg daily dexamethasone (or equivalent) for 7 days prior to start of treatment. Limited or occasional use of corticosteroids to treat or prevent acute adverse reactions is not considered an exclusion criterion.
25. Presence of active and uncontrolled infections or other severe concurrent disease, which, in the opinion of the investigator, would place the patient at undue risk or interfere with the study.
26. Concurrent malignancies unless the patient has been disease-free without intervention for at least 2 years.
27. Growth factors or immunomodulatory agents within 7 days prior to the administration of study treatment.
28. Serious, non-healing wound, ulcer, or bone fracture.
29. Requirement of concurrent therapy with anticoagulants at therapeutic doses.
30. Requirement of concurrent use of other anti-cancer treatments or agents other than study medication.
31. Any recent live vaccination within 4 weeks prior to treatment or plan to receive live vaccination during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of L19TNF plus lomustine with different administration sequences | From Day 1 to Day 42 of Cycle 1 (each cycle is 42 days)
  Occurrence of dose limiting toxicity (DLT) assessed by frequency and grade of adverse events (AE) according to CTCAE v.5.0.

SECONDARY OUTCOMES:
ORR | At 6 weeks, 12 weeks, 24 weeks and every 12 weeks up to 1 year
  Overall response rate
DCR | At 6 weeks, 12 weeks, 24 weeks and every 12 weeks through study completion, an average of 1 year
  Disease control rate
PFS | At 6 weeks, 12 weeks, 24 weeks and every 12 weeks through study completion, an average of 1 year
  Progression-free survival (PFS) based on iRANO criteria and a standardized MRI protocol
PFS at 6 months | At 6 months
  Progression-free survival (PFS) rate at 6 months
OS | At 6 weeks, 12 weeks, 24 weeks and every 12 weeks through study completion, an average of 1 year
  Overall survival (OS)
OS at 12 months | At 12 months
  Overall survival (OS) rate at 12 months
Safety (AE) | Throughout the study: from the enrolment through study completion, an average of 1 year
  Adverse events (AE) according to CTCAE v.5.0
Safety (SAE) | Throughout the study: from the enrolment through study completion, an average of 1 year
  Serious adverse events (SAE) according to CTCAE v.5.0
Safety (DILI) | Throughout the study: from the enrolment through study completion, an average of 1 year
  Drug induced liver injury (DILI) according to CTCAE v.5.0.

IPD SHARING:
Plan to Share IPD: No